CLINICAL TRIAL: NCT00269984
Title: A Double-Blind, Placebo-Controlled Study With Open-Label Follow-Up to Determine the Safety and Efficacy of r-HuEPO, Administered Subcutaneously, in Chronic Anemia Induced by Advanced Cancer
Brief Title: A Study to Determine the Safety and Effectiveness of Epoetin Alfa Versus Placebo in Patients With Persistent Anemia Caused by Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005833
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-04

CONDITIONS: Anemia
Keywords: Anemia; Blood transfusion; Epoetin alfa; Erythropoietin; Neoplasm; Epogen; Cancer
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin alfa

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of epoetin alfa versus placebo, injected beneath the skin, in the treatment of patients with persistent anemia caused by advanced cancer, with a below normal hematocrit of <= 37%. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production.

DETAILED DESCRIPTION:
Patients with advanced cancer frequently develop significant anemia, as determined by a blood test to measure hematocrit, with a below normal hematocrit of <=37%. Agents that can elevate the hematocrit level in patients with advanced cancer may increase the physical strength and stamina that is decreased by anemia, increase the patients' ability to persevere with chemotherapy, and improve their overall quality of life. Epoetin alfa is a genetically engineered form of a natural hormone, erythropoietin, that is used to treat anemia by stimulating red blood cell production. This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study to determine the safety and effectiveness of treatment with epoetin alfa in patients with persistent anemia caused by advanced cancer. Eligible patients will be randomly assigned to one of two treatment groups: epoetin alfa 100 units per kilogram or a comparable volume of placebo, given by injection beneath the skin. Patients will be given study medication 3 times weekly for up to 8 weeks or until a patient's hematocrit reaches 38% to 40%. The 8 weeks will be decreased to 4 weeks if, by Week 4, a patient's hematocrit decreases by more than 15% from the start of the study. At the end of the double-blind part of the study, patients who achieved a hematocrit level of 38 to 40%, or whose hematocrit decreased by >=15% from the start of the study by Week 4, will be allowed to enroll in the open-label part of the study for an additional 6 months and will receive epoetin alfa at a dose adjusted to maintain a hematocrit level between 38% and 40%. Within 5 to 7 days after it is documented that a patient's hematocrit has reached 38% to 40%, epoetin alfa will then be given once weekly by injection beneath the skin to maintain the hematocrit between 38% and 40% for the remaining time of the study. Patients will be seen by a healthcare professional once weekly and by the physician once monthly. Safety evaluations will include changes in laboratory tests, vital signs, physical examinations, electrocardiograms, and the incidence of adverse events from the start of the study to the end of the double-blind part of the study and to the end of the open-label part of the study. Effectiveness will be assessed by blood transfusion requirements and changes in hemoglobin, hematocrit, and immature red blood cell count from the start of the study to the end of study, as well as the physician's global evaluation and the quality of life assessment at the end of the double-blind part of the study and at the end of the open-label part of the study. The study hypothesis is that epoetin alfa will be well tolerated and more effective than placebo in stimulating adequate production of red blood cells in patients who are anemic as a result of advanced cancer. Double-blind: Epoetin alfa 100 units/kilogram (U/kg) or placebo injected under the skin; given 3 times weekly for 8 weeks or until hematocrit reaches 38%-40%. Open-label: Epoetin alfa 100 or 150 U/kg or a higher dose injected under the skin on a schedule to maintain hematocrit of 38%-40%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced cancer (except for rapid onset of severe leukemia and malignancies of the bone marrow and spleen) which is resistant to treatment or cure with chemotherapy or for which there is no established effective chemotherapy
* having persistent anemia as determined by a low hematocrit of <=37% and a negative direct Coombs' test (a blood test used to detect proteins and especially certain antibodies produced abnormally by some cancer cells on the surface of red blood cells)
* having a Performance score of 0, 1, 2, or 3 (patients' ability to perform daily activities, a score ranging from 0 [fully active, no disease restriction] to 3 [capable of only limited self-care, confined to bed or chair more than 50% of waking hours])
* having a life expectancy of at least 3 months
* who have not had chemotherapy to decrease cells and or radiation therapy within 1 month before the start of the study

Exclusion Criteria:

* Patients who have a history of any primary blood disease
* having signs and symptoms of significant disease/dysfunction not caused by the underlying cancer
* having an iron, folate, or vitamin B12 deficiency, or signs and symptoms suggestive of an autoimmune disease causing blood to break down and release iron-containing pigment
* having significant bleeding of the stomach and/or intestines, uncontrolled high blood pressure, a history of seizures, or a sudden onset of severe illness within 7 days before the start of the study
* received androgen therapy within 2 months before the start of the study or have used medications known to affect the hematocrit within 1 month before the start of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Study Completion 1990-06 (Actual)

PRIMARY OUTCOMES:
Changes in hemoglobin, hematocrit, and reticulocyte (immature red blood cells) count from before the study to the end of the study

SECONDARY OUTCOMES:
Safety assessment (laboratory tests, vital signs, adverse events, physical examination, electrocardiogram) from before study to end of double-blind study and to the end of open-label study; Physician's global evaluation; Quality of life assessment

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to determine the safety and effectiveness of epoetin alfa, injected beneath the skin, in patients with persistent anemia caused by advanced cancer — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=670&filename=CR005833_CSR.pdf